CLINICAL TRIAL: NCT07195929
Title: Blomia Tropicalis Allergen Extract. Determination of the Vivo Histamine Equivalent Prick Test Units
Brief Title: Determination of Blomia Tropicalis Allergen Extract in Prick Test Units
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M608-STD-067; 2024-515169-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Allergic Reactions; Allergic Skin Reaction
Keywords: Allergy; In-House Reference Preparation (IHRP); Prick test; Blomia tropicalis
MeSH Terms: conditions — Hypersensitivity | interventions — grass pollen extract, alum-adsorbed

STUDY DESIGN:
Intervention Model Description: Phase II trial, open-label, prospective, non-randomized, without a control group of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extract B. tropicalis + Positive control + Negative control (Experimental): There is only one treatment arm. In each subject, one drop of each of the three concentrations of both allergenic extracts, along with the positive (Histamine dihydrochloride 10 mg/mL) and negative (saline solution) controls, will be applied. Blomia tropicalis dilutions: 100 µg/mL and 20 µg/mL.
  Interventions: Other: Allergenic Extract

INTERVENTIONS:
Other: Allergenic Extract — In each subject, a drop of each of the 3 concentrations of the allergenic extract, in addition to the positive control (histamine) and the negative control, will be applied. The application will be duplicated on the subject's anterior forearm, with a distance of approximately 4 cm between each application to avoid overlapping reactions and false-positives results.
  Other Names: Allergenic Blomia tropicalis extract

SUMMARY:
The primary objective is to assess the concentration of Blomia tropicalis allergenic extract that induces a wheal of size equivalent to that produced by a 10 mg/mL histamine dihydrochloride solution, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
The trial will consist of a single visit, in which the following procedures will be carried out:

* Demographic data (age, race, and gender).
* Clinical history.
* Inclusion/exclusion criteria.
* Physical examination (cardiovascular, pulmonary, neurobiological, gastrointestinal, dermatological, other body systems and height, weight).
* Pregnancy test.
* Performance of prick-tests (3 concentrations of of Blomia tropicalis extract, positive control, and negative control).
* Collection of blood sample (10 mL) from the patient to create a pool of sera for in vitro standardization of the allergen extract.

Each serum sample will be labeled with the subject's number and frozen. These serum samples will remain in the freezer until the study concludes. Once the study is complete, they will be transported to the sponsor's facilities, where all sera will be pooled. This serum pool will be used for additional in vitro tests necessary to standardize and characterize the extract and produce its corresponding In-House Reference Product (IHRP), as indicated by the Spanish Pharmacopeia and the European Pharmacopeia. Additionally, it will be used in the necessary in vitro analyses for the standardization of new batches of the allergenic extract. After the serum pool is formed, the tubes containing the original serum samples are destroyed.

- Assessment of adverse events during the 72 hours following skin testing.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 to 64 years, both included.
2. Subjects who have signed and dated the informed consent form.
3. Subjects must reside in a geographical area where allergic problems caused by Blomia tropicalis are relevant.
4. Positive medical history of inhalant allergy (rhinitis and/or rhinoconjunctivitis and/or asthma) to Blomia tropicalis
5. A positive prick-test (mean wheal diameter ≥ 3 mm) with an extract of the same allergen and/or presence of specific IgE against complete extract or any molecular component to the allergenic source.
6. The area of the wheal obtained with 10 mg/mL histamine dihydrochloride should be ≥ 7 mm², which corresponds to a mean wheal diameter ≥ 3 mm.
7. The area of the wheal obtained with negative control should be < 7 mm², which corresponds to a mean wheal diameter < 3 mm.
8. Women of childbearing age (i.e following menarche and until postmenopause, defined as no menses for 12 months without an alternative medical cause, or non-subject to permanent sterilization methods, such as hysterectomy, bilateral salpingectomy and bilateral oophorectomy) must present a negative urine pregnancy test at the time of enrollment in the trial, as well as a confirmed menstrual period.
9. Women of childbearing age must commit to using a highly effective and adequate contraception method during the trial and up to 72 hours after the end of treatment with the investigational medicinal product. Such methods include combined (estrogen and progestogen containing) hormonal; contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence.

Exclusion Criteria:

1. Subjects outside the age range.
2. Subjects who have previously received immunotherapy within the last 5 years for the treatment of asthma or allergic rhinoconjunctivitis induced by allergens that may interfere with Blomia tropicalis extract.
3. Subjects with significant symptoms of rhinoconjunctivitis and/or bronchial asthma in whom discontinuation of systemic antihistamine treatment is contraindicated.
4. Subjects who have previously exhibited a severe adverse reaction during diagnostic skin prick tests.
5. Subjects on treatment with ß-blockers.
6. Use of drugs that could interfere with skin prick test reactions (e.g., antihistamines) (See Section 5.2).
7. Clinically unstable subjects (acute asthma, febrile, etc.).
8. Subjects with active urticaria lesions, severe active dermographism, severe atopic dermatitis, sunburn, eczema, psoriasis lesions in the area where the prick test is performed (risk of false positives).
9. Subjects with active herpes simplex viral infection, or herpes varicella zoster in the area where the prick test is performed.
10. Subjects with any pathology in which the administration of adrenaline is contraindicated (hyperthyroidism, hypertension, heart disease, etc.).
11. States in which the subject is unable to offer cooperation and severe psychiatric disorders.
12. Pregnant or potentially pregnant women and breastfeeding women.
13. Subjects with known phenol allergy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Size of the induced papule on the skin | 15 minutes
  Size of the induced papule on the skin when applying each of the concentrations of the allergenic extracts and the positive (histamine) and negative controls, using the prick test.

SECONDARY OUTCOMES:
Adverse reactions | 30 minutes
  The secondary outcome is to assess the safety and tolerability of Blomia tropicalis extract. Mild side reactions such as pruritus, erythema, local oedema may occur during the diagnostic skin test by prick test. There is a risk, albeit rare and exceptional, of systemic reactions, sometimes severe (urticaria, asthma, anaphylactic shock) (28) (urticaria, asthma, anaphylactic shock, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: María Inmaculada Sánchez Machín, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

REFERENCES:
- [Background] Skin tests used in type I allergy testing Position paper. Sub-Committee on Skin Tests of the European Academy of Allergology and Clinical Immunology. Allergy. 1989;44(s10):11-59. No abstract available. PMID 2683837
- [Background] Casanovas M, Maranon F, Bel I. Comparison of skin-prick test assay and reverse enzyme immunoassay competition (REINA-C) for biological activity of allergens. Clin Exp Allergy. 1994 Feb;24(2):134-9. doi: 10.1111/j.1365-2222.1994.tb00209.x. PMID 8187028
- [Background] Pawankar R. Allergic diseases and asthma: a global public health concern and a call to action. World Allergy Organ J. 2014 May 19;7(1):12. doi: 10.1186/1939-4551-7-12. eCollection 2014. No abstract available. PMID 24940476